CLINICAL TRIAL: NCT03960970
Title: Azithromycin-based Extended-spectrum Prophylaxis in Scheduled Cesarean Deliveries
Brief Title: Two-drug Antibiotic Prophylaxis in Scheduled Cesarean Deliveries
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RWJ Barnabas Health at Jersey City Medical Center (Other)
Responsible Party: Principal Investigator, Tali Wajsfeld, Principal Investigador, RWJ Barnabas Health at Jersey City Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Prophylaxis Trial
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Endometritis; Cesarean Section; Infection; Wound Infection
Keywords: Cesarean Delivery; Endometritis; Wound Infection; Azithromycin; Antibiotic Prophylaxis
MeSH Terms: conditions — Endometritis; Infections; Wound Infection | interventions — Azithromycin; Cefoxitin

STUDY DESIGN:
Intervention Model Description: Pregnant patients admitted to Labor and Delivery unit between June 2019 and July 2020 will be randomized to received either standard prophylaxis or azithromycin and cephalosporin for preoperative prophylaxis after inclusion and exclusion criteria are met and informed consent for participation is signed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- One-drug Prophylaxis (Active Comparator): Mefoxin 2g IV, Piggyback, once
  Interventions: Drug: Mefoxin 2g
- Two-drug Prophylaxis (Experimental): Mefoxin 2g IV, Piggyback, once and Azithromycin 500mg IV, Piggyback, once
  Interventions: Drug: Azithromycin 500 mg; Drug: Mefoxin 2g

INTERVENTIONS:
Drug: Azithromycin 500 mg — Additional IV Azithromycin 500 mg to Standard Prophylaxis
  Arms: Two-drug Prophylaxis
Drug: Mefoxin 2g — Standard Prophylaxis
  Other Names: Cefoxitin

SUMMARY:
Cesarean deliveries are the most common surgical procedure performed in the United States. A significant decrease in cesarean delivery associated maternal morbidity has been achieved with preoperative prophylactic single-dose cephalosporin, widely used before skin incision. Also, on laboring patients and/or with rupture of membranes, several studies suggest that adding azithromycin to standard cephalosporin prophylaxis is cost-effective and reduces overall rates of endometritis, wound infection, readmission, use of antibiotics and serious maternal events. Azithromycin has effective coverage against Ureaplasma, associated with increased rates of endometritis. Although two-drug regimen has been suggested for laboring and/or patients that undergo cesarean delivery, no studies have investigated the potential benefits of two-drug regimen in non-laboring patients.

DETAILED DESCRIPTION:
Cesarean deliveries are the most common surgical procedure performed in the United States, and scheduled cesarean deliveries account for at least 40% of all cesarean deliveries every year. A significant decrease in cesarean delivery associated maternal morbidity has been achieved with preoperative prophylactic single-dose cephalosporin given within 60 minutes of skin incision. Also, on laboring patients and/or with rupture of membranes, several studies suggest that adding azithromycin to standard cephalosporin prophylaxis is not only cost-effective but reduces overall rates of endometritis and wound infection. Azithromycin provides effective coverage against Ureaplasma, commonly associated with increased rates of endometritis. Although two-drug regimen has been suggested for laboring and/or patients that undergo cesarean delivery, no studies have investigated the potential benefits of two-drug regimen in non-laboring patients. No increase in neonatal morbidity was noted with adjunctive azithromycin prophylaxis, including adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 18 years or older
* Women undergoing primary or repeat cesarean delivery
* Singleton gestation
* Gestational age greater than 34 weeks
* Pregnant patients undergoing scheduled cesarean delivery
* Intact membranes
* Non-laboring
* Signed informed consent

Exclusion Criteria:

* Maternal age < 18 years
* Multi-fetal gestation
* Known allergy to cephalosporin or azithromycin
* Patient unwilling or unable to provide consent
* Diagnosis of rupture of membranes
* Intraamniotic infection, or any other active bacterial infection (e.g. pyelonephritis, pneumonia, abscess) at time of randomization.
* Immunocompromising medical conditions: HIV positive with CD4 count below 200, chronic steroid use, current diagnosis of cancer and/or chemotherapy age use
* Emergent cesarean precluding consent or availability of study medication
* Need for hysterectomy at time of delivery
* Use of antibiotic in the 72 hours prior to admission, with exception to patient receiving antibiotics for GBS
* Inability to contact patient on postpartum period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2019-09-15 (Estimated); Primary Completion 2019-09-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Rates of Endometritis | Up to 6 weeks after delivery
  Presence of at least two of the following signs with no other recognized cause: fever (temperature of at least 38°C [100.4°F]), abdominal pain, uterine tenderness, or purulent drainage from the uterus.
Rates of Wound Infection | Up to 6 weeks after delivery
  Presence of either superficial or deep incisional surgical-site infection characterized by cellulitis or erythema and induration around the incision or purulent discharge from the incision site with or without fever and included necrotizing fasciitis. Wound hematoma, seroma, abscess or breakdown alone in the absence of the preceding signs did not constitute infection.

SECONDARY OUTCOMES:
Rates of Maternal Fever | Up to 6 weeks after delivery
  Temperature equal or greater than 100.4F
Rates of Maternal Postpartum Readmission or Unscheduled Visit | Up to 6 weeks after delivery
  Admission to hospital or unscheduled appointment in additional to regular 1-week and 6-week postpartum visit
Rates of Postpartum Antibiotic Use | Up to 6 weeks after delivery
  Antibiotic use for any reason including other infections such as UTI and sepsis.
Rates of Serious Adverse Events | Up to 6 weeks after delivery
  MICU admission, thromboembolic events, sepsis, maternal death

OTHER OUTCOMES:
Rates of Neonatal Intensive Care Unit (NICU) Admission | Up to 6 weeks after delivery
  Neonatal Intensive Care Unit (NICU) Admission rather than prematurity
Rates of Neonatal Readmission | Up to 6 weeks after delivery
  Hospital readmission within 6 weeks of birth

CONTACTS AND LOCATIONS:
Overall Officials: Tali Wajsfeld, MD, Principal Investigator — RWJ Barnabas Health at Jersey City Medical Center
Locations (1):
- Jersey City Medical Center, Jersey City, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tita ATN, Rouse DJ, Blackwell S, Saade GR, Spong CY, Andrews WW. Emerging concepts in antibiotic prophylaxis for cesarean delivery: a systematic review. Obstet Gynecol. 2009 Mar;113(3):675-682. doi: 10.1097/AOG.0b013e318197c3b6. PMID 19300334
- [Background] Andrews WW, Hauth JC, Cliver SP, Savage K, Goldenberg RL. Randomized clinical trial of extended spectrum antibiotic prophylaxis with coverage for Ureaplasma urealyticum to reduce post-cesarean delivery endometritis. Obstet Gynecol. 2003 Jun;101(6):1183-9. doi: 10.1016/s0029-7844(03)00016-4. PMID 12798523
- [Background] Boggess KA, Tita A, Jauk V, Saade G, Longo S, Clark EAS, Esplin S, Cleary K, Wapner R, Letson K, Owens M, Blackwell S, Beamon C, Szychowski JM, Andrews W; Cesarean Section Optimal Antibiotic Prophylaxis Trial Consortium. Risk Factors for Postcesarean Maternal Infection in a Trial of Extended-Spectrum Antibiotic Prophylaxis. Obstet Gynecol. 2017 Mar;129(3):481-485. doi: 10.1097/AOG.0000000000001899. PMID 28178058
- [Background] Tita AT, Szychowski JM, Boggess K, Saade G, Longo S, Clark E, Esplin S, Cleary K, Wapner R, Letson K, Owens M, Abramovici A, Ambalavanan N, Cutter G, Andrews W; C/SOAP Trial Consortium. Adjunctive Azithromycin Prophylaxis for Cesarean Delivery. N Engl J Med. 2016 Sep 29;375(13):1231-41. doi: 10.1056/NEJMoa1602044. PMID 27682034
- [Background] Andrews WW, Shah SR, Goldenberg RL, Cliver SP, Hauth JC, Cassell GH. Association of post-cesarean delivery endometritis with colonization of the chorioamnion by Ureaplasma urealyticum. Obstet Gynecol. 1995 Apr;85(4):509-14. doi: 10.1016/0029-7844(94)00436-H. PMID 7898825
- [Background] Harper LM, Kilgore M, Szychowski JM, Andrews WW, Tita ATN. Economic Evaluation of Adjunctive Azithromycin Prophylaxis for Cesarean Delivery. Obstet Gynecol. 2017 Aug;130(2):328-334. doi: 10.1097/AOG.0000000000002129. PMID 28697108
- [Background] Tita AT, Hauth JC, Grimes A, Owen J, Stamm AM, Andrews WW. Decreasing incidence of postcesarean endometritis with extended-spectrum antibiotic prophylaxis. Obstet Gynecol. 2008 Jan;111(1):51-6. doi: 10.1097/01.AOG.0000295868.43851.39. PMID 18165392
- [Background] ACOG Practice Bulletin No. 120: Use of prophylactic antibiotics in labor and delivery. Obstet Gynecol. 2011 Jun;117(6):1472-1483. doi: 10.1097/AOG.0b013e3182238c31. No abstract available. PMID 21606770
- [Background] Skeith AE, Niu B, Valent AM, Tuuli MG, Caughey AB. Adding Azithromycin to Cephalosporin for Cesarean Delivery Infection Prophylaxis: A Cost-Effectiveness Analysis. Obstet Gynecol. 2017 Dec;130(6):1279-1284. doi: 10.1097/AOG.0000000000002333. PMID 29112658
- [Background] Smith C, Egunsola O, Choonara I, Kotecha S, Jacqz-Aigrain E, Sammons H. Use and safety of azithromycin in neonates: a systematic review. BMJ Open. 2015 Dec 9;5(12):e008194. doi: 10.1136/bmjopen-2015-008194. PMID 26656010
- [Background] Sutton AL, Acosta EP, Larson KB, Kerstner-Wood CD, Tita AT, Biggio JR. Perinatal pharmacokinetics of azithromycin for cesarean prophylaxis. Am J Obstet Gynecol. 2015 Jun;212(6):812.e1-6. doi: 10.1016/j.ajog.2015.01.015. Epub 2015 Jan 13. PMID 25595580
- [Background] Smaill FM, Grivell RM. Antibiotic prophylaxis versus no prophylaxis for preventing infection after cesarean section. Cochrane Database Syst Rev. 2014 Oct 28;2014(10):CD007482. doi: 10.1002/14651858.CD007482.pub3. PMID 25350672